CLINICAL TRIAL: NCT02331602
Title: Comparison of Anti-inflammatory Effects of Rivaroxaban Versus Dabigatran in Patients With Non-valvular Atrial Fibrillation (RIVAL-AF Study) -Multicenter Randomized Study-
Brief Title: Anti-inflammatory Effects of Rivaroxaban Versus Dabigatran
Acronym: RIVAL-AF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yokohama City University Medical Center (Other)
Collaborators: Yokohama City University (Other)
Responsible Party: Principal Investigator, Kiyoshi Hibi, Associate Professor, Division of Cardiology, Yokohama City University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kimura5656
Record Dates: First submitted 2014-01-05; First posted 2015-01-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; anticoagulation; inflammation
MeSH Terms: conditions — Atrial Fibrillation; Inflammation | interventions — Rivaroxaban; Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rivaroxaban (Active Comparator): Patients are assigned to receive rivaroxaban 15mg once daily for 12 months according to a computer-generated randomization sequence at the central registration center. Patients with creatinine clearance 30-49 mL/min receive rivaroxaban 10mg once daily.
  Interventions: Drug: Rivaroxaban
- dabigatran (Active Comparator): Patients are assigned to receive dabigatran 150mg twice daily for 12 months according to a computer-generated randomization sequence at the central registration center. Patients at a high risk of bleeding receive dabigatran 110mg twice daily.
  Interventions: Drug: Dabigatran

INTERVENTIONS:
Drug: Rivaroxaban — Patients are assigned to receive rivaroxaban 15mg once daily for 12 months. Patients with creatinine clearance 30-49 mL/min receive rivaroxaban 10mg once daily.
  Other Names: Xarelto
  Arms: rivaroxaban
Drug: Dabigatran — Patients are assigned to receive dabigatran 150mg twice daily for 12 months. Patients at a high risk of bleeding receive dabigatran 110mg twice daily.
  Other Names: Pradaxa
  Arms: dabigatran

SUMMARY:
The purpose of this study is to evaluate the antiinflammatory effects of rivaroxaban compared with dabigatran in patients with atrial fibrillation.

DETAILED DESCRIPTION:
Previous study showed that administration of rivaroxaban reduced expression of proinflammatory mediators in apolipoprotein E-deficient mice. However, it is unknown whether the anti-inflammatory markers are decreased in patients with atrial fibrillation receiving novel oral anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

* non-valvular atrial fibrillation
* a CHADS2-VASc score of 1 or more

Exclusion Criteria:

* contraindication for rivaroxaban or dabigatran
* stroke or systemic embolism, acute coronary syndromes or peripheral artery disease within 6 months before enrollment
* acute heart failure
* severe chronic renal failure (creatinine clearance < 30mL/min.)
* receiving dual antiplatelet therapy
* patients with a body weight of 50kg or less
* uncontrolled hypertension
* active malignancy, collagen disease, or infectious disease
* patients undergoing surgery within 6 months before enrollment
* patients who are planned to undergoing catheter ablation for atrial fibrillation
* patients who are not allowed to participate in the trial by judgement of the treating physician

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
median variation of inflammatory markers (including high sensitivity C reactive protein, pentraxin3, interleukin-6, and interleukin-18) between at baseline and 12 months later in each treatment group | 12 months

SECONDARY OUTCOMES:
change over time of above inflammatory markers during 12 months follow-up period (at baseline, 1 month, 3 months, 6 months, and 12 months later) in each treatment group | 12 months

OTHER OUTCOMES:
frequency of 12-month adverse cardiac and cerebrovascular events (including cardiovascular death, myocardial infarction, revascularization, ischemic stroke and systemic embolism)and frequency of 12-month major bleeding (defined as ISTH criteria) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kazuo Kimura, MD, Principal Investigator — Yokohama City University Medical Center
Locations (16):
- Japan (16):
  - Ashigara Kami Hospital, Ashigaura, Kanagawa
  - Chigasaki Municipal Hospital, Chigasaki, Kanagawa
  - Fujisawa City Hospital, Fujisawa, Kanagawa
  - Fujisawa Shounandai Hospital, Fujisawa, Kanagawa
  - Hadano Red Cross Hospital, Hadano, Kanagawa
  - National Hospital Organization Sagamihara National Hospital, Sagamihara, Kanagawa
  - Nagatsuta kousei general hospital, Yokohama, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Saiseikai Yokohama City Southern Hospital, Yokohama, Kanagawa
  - Kanagawa Cardiovascular and Respiratory Disease Center, Yokohama, Kanagawa
  - Yokohama Seamen's Insurance Hospital, Yokohama, Kanagawa
  - International Goodwill Hospital, Yokohama, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Yokosuka City hospital, Yokosuka, Kanagawa
  - International University of Health and Welfare Atami Hospital, Atami, Shizuoka
  - Omori Red Cross Hospital, Ohta, Tokyo